CLINICAL TRIAL: NCT00545233
Title: A Randomized, Open-label Study of the Effect of PEGASYS ® Plus COPEGUS® With or Without Concomitant Pioglitazone (Actos®) on Early Viral Kinetics in Treatment-naive Patients With Chronic Hepatitis C, Genotype-1, and Insulin Resistance
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) Plus COPEGUS (Ribavirin) With or Without Pioglitazone in Treatment-Naive Patients With Chronic Hepatitis C and Insulin Resistance.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21301
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin; Pioglitazone

ARMS (2):
- PEG-INF alpha-2a + ribavirin+ pioglitazone (Experimental): Participants received pioglitazone in a 16 week run-in period (30 mg per day orally for 8 weeks followed by 45 mg per day orally for 8 weeks). Participants then received piogliatzone 45 mg daily orally plus 18 μg of Peginterferon Alfa-2a (PEG-INF alpha-2a) subcutaneous (sc) once a week plus ribavirin (1000 - 1600 mg/day orally as a split dose in the morning and the evening based on the participant's body weight) for 48 weeks in the anti-HCV treatment phase. Participants received 45 mg of pioglitazone per day orally in the 24 week follow-up period.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]; Drug: Pioglitazone
- PEG-INF alpha-2a + ribavirin (Active Comparator): Participants received 18 μg of Peginterferon Alfa-2a (PEG-INF alpha-2a) subcutaneous (sc) once a week plus ribavirin (1000 - 1600 mg/day orally as a split dose in the morning and the evening based on the participant's body weight) for 48 weeks in the anti-HCV treatment phase followed by a treatment free 24 week follow-up period.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms subcutaneous weekly for 48 weeks
  Other Names: Pegasys
Drug: ribavirin [Copegus] — 1000-1600 mg day orally for 48 weeks.
  Other Names: Copegus
Drug: Pioglitazone — 30 mg daily for 8 weeks increasing to 45 mg daily for 64 weeks.
  Other Names: Actos
  Arms: PEG-INF alpha-2a + ribavirin+ pioglitazone

SUMMARY:
This 2 arm study will assess the efficacy and safety of PEGASYS plus COPEGUS, with or without concomitant pioglitazone, on hepatitis C virus titers in treatment-naive patients with genotype 1 chronic hepatitis C, and insulin resistance. Patients will be randomized to receive either a)PEGASYS 180 micrograms/week + Copegus 1000-1600 mg/day (according to body weight) for 48 weeks or b)16 weeks of pioglitazone (30 mg daily for 8 weeks, then 45 mg daily for 8 weeks), followed by PEGASYS 180 micrograms/week + Copegus 1000-1600 mg/day + pioglitazone 45 mg daily for 48 weeks. The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic hepatitis C, genotype 1;
* insulin resistance.

Exclusion Criteria:

* other forms of liver disease;
* cirrhosis;
* previous treatment for chronic hepatitis C;
* insulin treatment during prior 2 weeks;
* type 1 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (57):
- United States (56):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Anaheim, California
  - Fresno, California
  - La Jolla, California
  - Loma Linda, California
  - Los Angeles, California
  - Merced, California
  - Palo Alto, California
  - Pasadena, California
  - San Clemente, California
  - San Mateo, California
  - Englewood, Colorado
  - Littleton, Colorado
  - Hartford, Connecticut
  - Atlanta, Georgia
  - Chicago, Illinois
  - Downers Grove, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Duluth, Minnesota
  - Tupelo, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Egg Harbour Township, New Jersey
  - Hackensack, New Jersey
  - Bayside, New York
  - Manhasset, New York
  - New York, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - West Nashville, Tennessee
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Tacoma, Washington
- San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients randomized to the pioglitazone arm participated in a 16-week pioglitazone run-in (Week -16 to Week 0) prior to beginning anti-HCV therapy: PEG-INF alpha-2a [Pegasys] plus ribavarin [Copegus]. Patients randomized to the without pioglitazone arm started anti-HCV therapy immediately.
Groups:
- PEG-INF Alpha-2a + Ribavirin+ Pioglitazone: Participants received pioglitazone in a 16 week run-in period (30 mg per day orally for 8 weeks followed by 45 mg per day orally for 8 weeks). Participants then received pioglitazone 45 mg daily orally plus 18 μg of Peginterferon Alfa-2a (PEG-INF alpha-2a)[Pegasys] subcutaneous (sc) once a week plus ribavirin [Copegus] (1000 - 1600 mg/day orally as a split dose in the morning and the evening based on the participant's body weight) for 48 weeks in the anti-HCV treatment phase. Participants received 45 mg of pioglitazone per day orally in the 24 week follow-up period.
- PEG-INF Alpha-2a + Ribavirin: Participants received 18 μg of Peginterferon Alfa-2a (PEG-INF alpha-2a)[Pegasys] subcutaneous (sc) once a week plus ribavirin [Copegus] (1000 - 1600 mg/day orally as a split dose in the morning and the evening based on the participant's body weight) for 48 weeks in the anti-HCV treatment phase followed by a treatment free 24 week follow-up period.
Period: Overall Study
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Started | 79 | 76
Safety Set | 77 | 75
Intent-to-Treat (ITT) | 77 | 73
Completed | 33 | 41
Not Completed | 46 | 35
Not completed — Adverse Event | 10 | 5
Not completed — Violation of Selection Criteria at Entry | 5 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Refused Treatment | 9 | 7
Not completed — Failure to Return | 4 | 6
Not completed — Insufficient response | 14 | 15
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin | Total
Number analyzed (Participants) | 77 | 73 | 150
Age, Customized [Number; unit: participants] — Baseline Measures are based on the Intent-to-Treat Population that includes all participants who received at least one dose of study drug.
  participants
    <=40 years | 6 | 8 | 14
    >40 years | 71 | 65 | 136
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 50 | 45 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change From Initiation of Pegasys Plus Copegus in log10 Hepatitis C Virus Ribonucleic Acid (HCV RNA) Viral Load to Week 12 of Anti-HCV Therapy
Description: Serum samples were collected for HCV RNA. The change from initiation of Pegasys plus Copegus to Week 12 in HCV RNA titers were calculated. Randomization for the with Pioglitazone arm occurred prior to the 16 week run-in period and randomization for the without Pioglitazone arm occurred prior to the start of anti-HCV treatment.
Time Frame: Initiation of Pegasys plus Copegus, Week 12 of anti-HCV treatment
Population: Intent-to Treat population includes all randomized patients who received at least one dose of study drug and had at least one post-randomization HCV RNA assessment. Last Observation Carried Forward (LOCF) was used to replace missing data after dropout with the last observed data.
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
IU/mL | -3.5 (0.22) | -3.7 (0.19)

2. Secondary Outcome: Change From Initiation of Pegasys Plus Copegus in log10 HCV RNA Viral Load to Week 24 and Week 48 of Anti-HCV Therapy
Description: Serum samples were collected for HCV RNA. The change from Initiation of Pegasys Plus Copegus to Week 24 and Week 48 in HCV RNA titers were calculated. Randomization for the with Pioglitazone arm occurred prior to the 16 week run-in period and randomization for the without Pioglitazone arm occurred prior to the start of anti-HCV treatment.
Time Frame: Initiation of Pegasys Plus Copegus, Week 24 and Week 48 of anti-HCV therapy
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
IU/mL
  Week 24 (N=60, 72) | -4.0 (0.23) | -3.9 (0.21)
  Week 48 (N=62, 73) | -3.5 (0.27) | -3.6 (0.24)

3. Secondary Outcome: Percentage of Participants Achieving Virologic Response
Description: Virologic response was defined as undetectable HCV RNA < 28 IU/mL. Patients with missing HCV RNA values are considered as non-responders.
Time Frame: Weeks 4, 12, 24, 48, 60, 72
Population: Intent-to Treat population includes all randomized patients who received at least one dose of study drug and had at least one post-randomization HCV RNA assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
Percentage of Participants
  Weeks 4 | 6.5 | 16.4
  Week 12 | 33.8 | 49.3
  Week 24 | 46.8 | 63.0
  Week 48 | 39.0 | 56.2
  Week 60 | 26.0 | 39.7
  Week 72 | 26.0 | 38.4

4. Secondary Outcome: Percentage of Participants With a ≥ 2 log10 Decrease in HCV RNA From Initiation of Pegasys Plus Copegus to Weeks 4, 12, 24, 48, 60, 72
Description: Serum samples were collected for HCV RNA. The percentage of participants with a ≥ 2 log10 decrease in HCV RNA from initiation of Pegasys plus Copegus to time point was calculated.
Time Frame: Initiation of Pegasys plus Copegus, Weeks 4, 12, 24, 48, 60, 72
Population: Intent-to Treat population included all randomized patients who received at least one dose of study drug and had at least one post-randomization HCV RNA assessment. Patients with missing HCV RNA values are considered as non-responders.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
Percentage of Participants
  Weeks 4 | 41.6 | 52.1
  Week 12 | 58.4 | 76.7
  Week 24 | 51.9 | 72.6
  Week 48 | 39.0 | 54.8
  Week 60 | 26.0 | 41.1
  Week 72 | 26.0 | 37.0

5. Secondary Outcome: Percentage of Participants With a Virological Relapse at Week 72 (24 Weeks After the End of Anti-HCV Treatment)
Description: Virologic relapse was defined as the reappearance of HCV-RNA in serum after PEG-INF alpha 2a therapy is discontinued in a patient who was HCV-RNA undetectable at the completion of anti-HCV therapy.
Time Frame: Week 72
Population: Intent-to Treat population includes all randomized patients who received at least one dose of study drug and had at least one post-randomization HCV RNA assessment. Patients with missing HCV RNA values are considered as non-responders.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
Percentage of Participants | 15.6 | 19.2

6. Secondary Outcome: Percentage of Participants With a Confirmed Virological Breakthrough up to 48 Weeks
Description: Virological breakthrough is a detectable HCV RNA at any time during anti-HCV treatment up to Week 48 after the attainment of undetectable HCV RNA.
Time Frame: Up to 48 Weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
Percentage of Participants | 15.6 | 13.7

7. Secondary Outcome: Percentage of Nonresponders During the 48 Week Anti-HCV Treatment Period
Description: Nonresponders are defined as patients who did not achieve undetectable HCV RNA during anti-HCV treatment
Time Frame: Up to 48 Weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
Percentage of Participants | 45.5 | 30.1

8. Secondary Outcome: Change in Log10 HCV RNA Viral Load at Assessments From Randomization to 16 Weeks of Pioglitazone Pretreatment Run-In Period for the Pioglitazone Arm Only
Description: Serum HCV RNA was collected at randomization and during the pioglitazone run-in period at various time points for the with pioglitazone arm only. The change from randomization to each of these time points was calculated.
Time Frame: Randomization (Week-16),Weeks -12, -8, -4 and 0
Population: as for outcome 5
Measure: Mean (Standard Error); unit: IU/mL
Groups:
- PEG-INF Alpha-2a + Ribavirin+ Pioglitazone: Participants received pioglitazone in a 16 week run-in period (30 mg per day orally for 8 weeks followed by 45 mg per day orally for 8 weeks). Participants then received piogliatzone 45 mg daily orally plus 18 μg of Peginterferon Alfa-2a (PEG-INF alpha-2a) subcutaneous (sc) once a week plus ribavirin (1000 - 1600 mg/day orally as a split dose in the morning and the evening based on the participant's body weight) for 48 weeks in the anti-HCV treatment phase. Participants received 45 mg of piogliatzone per day orally in the 24 week follow-up period.
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone
Number analyzed (Participants) | 77
IU/mL
  Week -12 (n=74) | -0.01 (0.037)
  Week -8 (n=68) | 0.00 (0.049)
  Week -4 (n=66) | 0.07 (0.048)
  Week 0 (n=64) | -0.03 (0.046)

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Levels at Each Time Point Assessed
Description: Blood was collected for plasma fasting glucose levels at various time points throughout the study and was used as a measure of glycemic control (monitoring the ability of the patient to maintain normal blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: Participants from the Intent-to Treat population who received at least one dose of study drug and who had data available at the given time point for analysis.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
mmol/L
  Week 4 (n=58, 70) | -0.4 (0.24) | -0.2 (0.17)
  Week 8 (n=57, 68) | -0.7 (0.25) | -0.1 (0.33)
  Week 12 (n=55, 66) | -0.8 (0.25) | -0.6 (0.28)
  Week 16 (n=53, 61) | -0.8 (0.26) | -0.5 (0.36)
  Week 20 (n=46, 57) | -0.6 (0.19) | -0.3 (0.19)
  Week 24 (n=47, 61) | -0.5 (0.30) | -0.3 (0.15)
  Week 28 (n=51, 62) | -0.4 (0.16) | -0.3 (0.16)
  Week 32 (n=39, 47) | -0.5 (0.19) | -0.5 (0.23)
  Week 36 (n=38, 46) | -0.6 (0.20) | -0.4 (0.23)
  Week 40 (n=44, 50) | -0.4 (0.20) | -0.7 (0.20)
  Week 44 (n=37, 43) | -0.4 (0.33) | -0.2 (0.25)
  Week 48 (n=34, 46) | -0.5 (0.22) | -0.1 (0.24)
  Week 60 (n=33, 41) | -0.6 (0.23) | -0.1 (0.34)
  Week 72 (n=30, 38) | -0.6 (0.22) | -0.1 (0.31)

10. Secondary Outcome: Change From Baseline in Fasting Insulin Levels at Each Time Point Assessed.
Description: Blood was collected for fasting insulin levels at various time points throughout the study and was used as a measure of glycemic control (monitoring the ability of the patient to maintain normal blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
pmol/L
  Week 4 (N=56, 43) | 6.4 (20.9) | -28.4 (30.1)
  Week 8 (N=4, 27) | -40.6 (33.1) | 7.3 (37.1)
  Week 12 (N=52, 65) | -34.4 (17.2) | -36.0 (23.8)
  Week 16 (N=5, 5) | -59.0 (49.9) | -162.2 (198.8)
  Week 20 (N=2, 3) | 132.6 (127.8) | 180.1 (644.4)
  Week 24 (N=42, 60) | -38.4 (16.7) | -29.1 (10.1)
  Week 28 (N=12, 13) | 11.8 (44.6) | -21.2 (30.1)
  Week 32 (N=2, 3) | -47.2 (36.8) | 41.7 (119.5)
  Week 36 (N=0, 2) | NA (NA) — No participants with data in this arm at Week 36. | 41.0 (33.3)
  Week 40 (N=8, 2) | 2.0 (71.0) | 62.2 (76.0)
  Week 44 (N=4, 0) | 370.5 (405.6) | NA (NA) — No participants with data for this arm at Week 44.
  Week 48 (N=32, 46) | -38.0 (20.7) | -14.3 (17.2)
  Week 60 (N=1, 3) | -13.2 (NA) — Only 1 participant with data. Unable to calculate standard error. | 91.0 (66.8)
  Week 72 (N=30, 40) | -61.4 (17.2) | -4.8 (26.3)

11. Secondary Outcome: Change From Baseline in Fasting Hemoglobin A1C (HbA1c) Concentrations at Each Time Point Assessed
Description: Blood was collected for a fasting Hemoglobin A1C level at various time points throughout the study and was used as a measure of glycemic control (monitoring the ability of the patient to maintain normal blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Percent
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
Percent
  Week 4 (n=3, 5) | -0.4 (0.35) | -0.1 (0.22)
  Week 8 (n=4, 28) | -0.9 (0.13) | -1.0 (0.18)
  Week 12 (n=50, 65) | -1.1 (0.10) | -1.5 (0.12)
  Week 16 (n=5, 4) | -0.8 (0.12) | -1.7 (0.64)
  Week 20 (n=1, 4) | -0.6 (NA) — Only 1 participant unable to calculate standard error. | -1.3 (0.30)
  Week 24 (n=41, 51) | -1.0 (0.10) | -1.5 (0.12)
  Week 28 (n=11, 12) | -0.7 (0.20) | -1.1 (0.17)
  Week 32 (n=2, 2) | -1.0 (0.40) | -1.7 (0.80)
  Week 36 (n=0, 2) | NA (NA) — No participants with data in this arm for Week 36. | -0.5 (0.05)
  Week 40 (n=8, 1) | -0.3 (0.28) | -1.8 (NA) — Only 1 participant with data. Unable to calculate standard error.
  Week 44 (n=7, 0) | -0.7 (0.22) | NA (NA) — No participants with data in this arm at Week 44.
  Week 48 (N=31, 46) | -0.8 (0.13) | -1.1 (0.15)
  Week 60 (N=1, 2) | -0.2 (NA) — Only 1 participant with data. Unable to calculate standard error. | -0.1 (0.30)
  Week 72 (N=29, 38) | -0.1 (0.10) | -0.1 (0.11)

12. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment (HOMA) Scores at Each Time Point Assessed
Description: Insulin resistance (IR) is calculated using the following formula:
  HOMA score = (fasting glucose in mg/dL × fasting insulin in μIU/mL) / 405.
  Baseline for "with pioglitazone" arm occurred prior to the start of 16 week run-in period and for "without pioglitazone" arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the start of anti-HCV therapy is calculated.
  A normal patient can have a HOMA score up to 3. A patient with a score of >3 is definitely IR. Patients scoring 2-3 can be IR but other factors may be causing this without being IR.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: HOMA Score
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
HOMA Score
  Week 4 (n=54, 42) | 0.6 (1.31) | -0.8 (1.52)
  Week 8 (n=3, 25) | -2.3 (1.74) | 0.6 (1.80)
  Week 12 (n=51, 63) | -2.0 (0.74) | -2.1 (1.07)
  Week 16 (n=5, 5) | -3.2 (2.28) | -9.1 (7.96)
  Week 20 (n=2, 3) | 4.0 (4.60) | 10.5 (32.38)
  Week 24 (n=42, 60) | -1.8 (0.74) | -1.3 (0.45)
  Week 28 (n=10, 13) | 0.8 (1.95) | -1.0 (1.36)
  Week 32 (n=2, 2) | -1.8 (1.27) | 4.2 (6.81)
  Week 36 (n=0, 2) | NA (NA) — No participants with data in this arm at Week 36. | 2.0 (0.41)
  Week 40 (n=6, 2) | 0.2 (4.00) | 1.0 (3.91)
  Week 44 (n=4, 0) | 30.4 (31.74) | NA (NA) — No participants with data in this arm at Week 44.
  Week 48 (n=30, 44) | -1.6 (0.98) | -0.3 (0.91)
  Week 60 (n=1, 2) | 0.6 (NA) — Only 1 participant with data. Unable to calculate standard error. | 5.0 (3.83)
  Week 72 (n=27, 35) | -2.7 (1.01) | -0.1 (1.39)

13. Secondary Outcome: Change From Baseline in Serum Triglyceride Concentrations at Each Time-point Assessed
Description: Blood was collected and assayed for fasting serum triglyceride levels at various time points throughout the study and was used as an indicator of lipid control.
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60, 72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
mmol/L
  Week 4 (n=61, 72) | 0.5 (0.21) | 0.4 (0.11)
  Week 8 (n=58, 69) | 0.2 (0.09) | 0.5 (0.12)
  Week 12 (n=56, 68) | 0.2 (0.11) | 0.7 (0.23)
  Week 16 (n=53, 62) | 0.2 (0.08) | 0.6 (0.20)
  Week 20 (n=46, 59) | 0.2 (0.11) | 0.6 (0.16)
  Week 24 (n=47, 61) | 0.5 (0.26) | 0.3 (0.10)
  Week 28 (n=52, 62) | 0.2 (0.10) | 0.4 (0.14)
  Week 32 (n=38, 47) | 0.3 (0.13) | 0.5 (0.19)
  Week 36 (n=38, 46) | 0.1 (0.11) | 0.5 (0.15)
  Week 40 (n=45, 49) | 0.2 (0.12) | 0.4 (0.13)
  Week 44 (n=37, 43) | 0.3 (0.23) | 0.3 (0.12)
  Week 48 (n=34, 46) | 0.2 (0.13) | 0.5 (0.18)
  Week 60 (n=33, 41) | -0.2 (0.11) | 0.3 (0.16)
  Week 72 (n=30, 39) | -0.1 (0.16) | 0.2 (0.12)

14. Secondary Outcome: Change From Baseline in Total Cholesterol Levels at Each Time-point Assessed
Description: Blood was collected and assayed for fasting serum cholesterol levels at various time points throughout the study and was used as an indicator of lipid control.
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
mmol/L
  Week 4 (n=61, 72) | -0.2 (0.08) | -0.5 (0.07)
  Week 8 (n=58, 69) | -0.2 (0.07) | -0.6 (0.08)
  Week 12 (n=56, 68) | -0.2 (0.07) | -0.6 (0.09)
  Week 16 (n=53, 62) | -0.3 (0.07) | -0.7 (0.11)
  Week 20 (n=46, 59) | -0.3 (0.08) | -0.6 (0.11)
  Week 24 (n=47, 61) | -0.2 (0.09) | -0.7 (0.10)
  Week 28 (n=52, 62) | -0.3 (0.08) | -0.7 (0.10)
  Week 32 (n=38, 47) | -0.4 (0.10) | -0.8 (0.11)
  Week 36 (n=38, 46) | -0.3 (0.10) | -0.7 (0.12)
  Week 40 (n=45, 49) | -0.3 (0.08) | -0.8 (0.12)
  Week 44 (n=37, 43) | -0.2 (0.11) | -0.8 (0.13)
  Week 48 (n=34, 46) | -0.3 (0.11) | -0.7 (0.11)
  Week 60 (n=33, 41) | 0.0 (0.15) | 0.1 (0.14)
  Week 72 (n=30, 39) | 0.3 (0.15) | 0.2 (0.14)

15. Secondary Outcome: Change From Baseline in Low-density Lipoprotein (LDL-cholesterol) Levels at Each Time-point Assessed
Description: Blood was collected and assayed for fasting serum low-density lipoprotein (LDL-cholesterol) levels at various time points throughout the study and was used as an indicator of lipid control.
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
mmol/L
  Week 4 (n=58, 70) | -0.3 (0.07) | -0.5 (0.07)
  Week 8 (n=57, 66) | -0.2 (0.06) | -0.6 (0.08)
  Week 12 (n=55, 62) | -0.2 (0.07) | -0.5 (0.10)
  Week 16 (n=53, 58) | -0.2 (0.07) | -0.6 (0.10)
  Week 20 (n=46, 56) | -0.2 (0.07) | -0.6 (0.11)
  Week 24 (n=45, 60) | -0.2 (0.08) | -0.6 (0.10)
  Week 28 (n=52, 60) | -0.2 (0.08) | -0.6 (0.09)
  Week 32 (N=38, 44) | -0.40 (0.09) | -0.7 (0.12)
  Week 36 (n=37, 44) | -0.2 (0.08) | -0.7 (0.11)
  Week 40 (n=44, 49) | -0.3 (0.08) | -0.7 (0.11)
  Week 44 (n=36, 43) | -0.2 (0.08) | -0.7 (0.11)
  Week 48 (n=34, 44) | -0.3 (0.09) | -0.7 (0.10)
  Week 60 (n=33, 39) | 0.1 (0.12) | 0.1 (0.13)
  Week 72 (n=30, 38) | 0.2 (0.10) | 0.0 (0.13)

16. Secondary Outcome: Change From Baseline in High-density Lipoprotein (HDL-cholesterol) Levels at Each Time-point Assessed
Description: Blood was collected and assayed for fasting high-density lipoprotein (HDL-cholesterol) levels at various time points throughout the study and was used as an indicator of lipid control.
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4,8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
mmol/L
  Week 4 (n=61, 72) | -0.1 (0.04) | -0.1 (0.03)
  Week 8 (n=58, 69) | -0.1 (0.03) | -0.2 (0.03)
  Week 12 (n=56, 68) | -0.1 (0.03) | -0.2 (0.03)
  Week 16 (n=53, 62) | -0.2 (0.03) | -0.2 (0.03)
  Week 20 (n=46, 59) | -0.1 (0.04) | -0.2 (0.04)
  Week 24 (n=47, 61) | -0.2 (0.03) | -0.2 (0.04)
  Week 28 (n=52, 62) | -0.1 (0.03) | -0.2 (0.04)
  Week 32 (n=38, 47) | -0.2 (0.04) | -0.3 (0.04)
  Week 36 (n=38, 46) | -0.1 (0.04) | -0.3 (0.05)
  Week 40 (n=45, 49) | -0.1 (0.03) | -0.3 (0.05)
  Week 44 (n=37, 43) | -0.1 (0.04) | -0.2 (0.05)
  Week 48 (n=34, 46) | -0.1 (0.05) | -0.2 (0.05)
  Week 60 (n=33, 41) | 0.1 (0.06) | -0.1 (0.04)
  Week 72 (n=30, 39) | 0.2 (0.07) | 0.1 (0.04)

17. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor Alpha (TNF-α) at Each Time Point Assessed
Description: Blood was collected for tumor necrosis factor alpha at various time points throughout the study and was used as a measure of insulin resistance (the inability of insulin to control blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
pg/mL
  Week 4 (n=56, 41) | -1.9 (0.88) | -0.9 (1.26)
  Week 8 (n=5, 25) | -3.7 (3.93) | 1.1 (0.36)
  Week 12 (n=51, 45) | -2.0 (0.89) | 2.8 (3.84)
  Week 16 (n=5, 4) | -1.2 (1.74) | 0.6 (1.85)
  Week 20 (n=2, 3) | 0.7 (0.38) | -3.5 (3.64)
  Week 24 (n=42, 57) | -1.1 (1.50) | -1.8 (1.31)
  Week 28 (n=12, 12) | -0.7 (1.73) | -0.1 (0.68)
  Week 32 (n=2, 2) | -0.8 (0.90) | -1.0 (0.07)
  Week 36 (n=0, 2) | NA (NA) — No participants with data in this arm for Week 36 | 2.7 (2.66)
  Week 40 (n=7, 1) | -3.3 (1.58) | 3.6 (NA) — Only 1 participant unable to calculate standard error
  Week 44 (n=4, 0) | -2.1 (0.35) | NA (NA) — No participants with data in this arm for Week 44
  Week 48 (n=32, 44) | -2.5 (0.91) | -1.4 (1.33)
  Week 60 (n=1, 2) | -2.4 (NA) — Only 1 participant unable to calculate standard error | -1.4 (0.20)
  Week 72 (n=29, 37) | -3.7 (1.54) | -2.0 (0.31)

18. Secondary Outcome: Change From Baseline in Transforming Growth Factor Beta (TGF-β) Levels at Each Time Point Assessed
Description: Blood was collected for Transforming Growth Factor beta at various time points throughout the study and was used as a measure of insulin resistance (the inability of insulin to control blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
pg/mL
  Week 4 (n=56, 41) | -14891 (1406) | -7256 (1711)
  Week 8 (n=5, 25) | -16224 (8318) | -13955 (2190)
  Week 12 (n=51, 45) | -17666 (1655) | -11447 (2141)
  Week 16 (n=5, 4) | -6164 (8199) | -14570 (4272)
  Week 20 (n=2, 3) | -10653 (1886) | -11290 (10160)
  Week 24 (n=42, 57) | -15976 (1727) | -13875 (1619)
  Week 28 (n=12, 12) | -4071 (2864) | -9242 (3185)
  Week 32 (n=2, 2) | -19750 (12614) | -18973 (5737)
  Week 36 (n=0, 2) | NA (NA) — No participants with data in this arm for Week 36 | 8724 (12181)
  Week 40 (n=7, 1) | -3119 (4460) | 1785 (NA) — Only 1 participant unable to calculate standard error
  Week 44 (n=4, 0) | -6415 (5890) | NA (NA) — No participants with data in this arm for Week 44
  Week 48 (n=32, 44) | -16510 (2573) | -10149 (2285)
  Week 60 (n=1, 2) | -14539 (NA) — Only 1 participant unable to calculate standard error | -3612 (5410)
  Week 72 (n=29, 37) | -6403 (2504) | -1347 (2327)

19. Secondary Outcome: Change From Baseline in Adiponectin Levels at Each Time Point Assessed
Description: Blood was collected for adiponectin at various time points throughout the study and was used as a measure of insulin resistance (the inability of insulin to control blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: μg/mL
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
μg/mL
  Week 4 (n=56, 39) | 13.0 (1.15) | 1.6 (0.80)
  Week 8 (n=5, 23) | 12.2 (5.11) | -1.1 (0.60)
  Week 12 (n=49, 45) | 10.7 (1.17) | 0.3 (0.59)
  Week 16 (n=5, 4) | 9.0 (2.30) | -1.0 (0.41)
  Week 20 (n=2, 3) | 3.0 (2.00) | 4.0 (0.58)
  Week 24 (n=41, 55) | 12.5 (1.27) | 0.2 (0.57)
  Week 28 (n=11, 11) | 4.4 (2.18) | -1.0 (1.39)
  Week 32 (n=2, 2) | 13.0 (4.00) | 1.5 (0.50)
  Week 36 (n=0, 2) | NA (NA) — No participants with data in this arm for Week 36 | 0.0 (1.00)
  Week 40 (n=7, 1) | 2.9 (1.61) | -4.0 (NA) — Only 1 participant unable to calculate standard error
  Week 44 (n=3, 0) | 3.7 (1.67) | NA (NA) — No participants with data in this arm for Week 44
  Week 48 (n=31, 44) | 10.8 (1.70) | 0.3 (0.62)
  Week 60 (n=1, 2) | -1.0 (NA) — Only 1 participant unable to calculate standard error | 3.0 (1.00)
  Week 72 (n=29, 36) | 8.2 (2.07) | -0.1 (0.38)

20. Secondary Outcome: Change From Baseline in Leptin Levels at Each Time Point Assessed
Description: Blood was collected for leptin at various time points throughout the study and was used as a measure of insulin resistance (the inability of insulin to control blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
ng/mL
  Week 4 (n=56, 39) | -1.8 (1.38) | -2.4 (0.73)
  Week 8 (n=5, 22) | -1.9 (1.43) | -3.0 (0.89)
  Week 12 (n=48, 44) | -3.1 (1.38) | -3.8 (1.01)
  Week 16 (n=5, 4) | -6.4 (6.67) | -7.9 (7.37)
  Week 20 (n=2, 3) | -2.9 (0.70) | -4.0 (1.85)
  Week 24 (n=42, 54) | -5.8 (1.55) | -5.0 (0.84)
  Week 28 (n=11, 11) | -3.7 (2.05) | -4.1 (1.93)
  Week 32 (n=2, 2) | -4.5 (1.10) | -4.9 (0.90)
  Week 36 (n=0, 2) | NA (NA) — No participants with data in this arm for Week 36 | -1.5 (1.20)
  Week 40 (n=7, 1) | -4.8 (2.32) | 11.5 (NA) — Only 1 participant unable to calculate standard error
  Week 44 (n=3, 0) | 6.0 (8.70) | NA (NA) — No participants with data in this arm for Week 44
  Week 48 (n=31, 43) | -4.6 (1.31) | -5.5 (1.25)
  Week 60 (n=1, 2) | 3.4 (NA) — Only 1 participant unable to calculate standard error | -0.6 (1.50)
  Week 72 (n=29, 36) | 1.3 (2.12) | 1.4 (1.17)

21. Secondary Outcome: Change From Baseline in Free Fatty Acid Levels at Each Time Point Assessed
Description: Blood was collected for free fatty acids at various time points throughout the study and was used as a measure of insulin resistance (the inability of insulin to control blood sugar levels).
  Baseline for the with pioglitazone arm occurred prior to the start of 16 week run-in period and for the without pioglitazone arm prior to the start of anti-HCV therapy. The change from baseline to Weeks 4 thru 72 after the initiation of anti-HCV therapy is calculated.
Time Frame: Baseline, Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 73
mmol/L
  Week 4 (n=55, 35) | 0.0 (0.09) | 0.1 (0.05)
  Week 8 (n=2, 2) | -0.1 (0.08) | 0.0 (0.31)
  Week 12 (n=52, 32) | -0.0 (0.07) | 0.2 (0.12)
  Week 16 (n=5, 3) | -0.0 (0.16) | -0.1 (0.26)
  Week 20 (n=2, 3) | -0.5 (0.34) | 0.1 (0.38)
  Week 24 (n=40, 31) | -0.1 (0.09) | 0.2 (0.05)
  Week 28 (n=11, 5) | 0.0 (0.09) | 0.1 (0.13)
  Week 32 (n=2, 1) | 0.3 (0.12) | -0.4 (NA) — Only 1 participant unable to calculate standard error
  Week 36 (n=0, 1) | NA (NA) — No participants with data in this arm for Week 36 | 0.2 (NA) — Only 1 participant unable to calculate standard error
  Week 40 (n=8, 1) | 0.2 (0.31) | -0.3 (NA) — Only 1 participant unable to calculate standard error
  Week 44 (n=4, 0) | -0.0 (0.05) | NA (NA) — No participants with data in this arm for Week 44
  Week 48 (n=32, 24) | -0.2 (0.09) | 0.0 (0.05)
  Week 60 (n=1, 0) | 0.1 (NA) — Only 1 participant unable to calculate standard error | NA (NA) — No participants with data in this arm for Week 60
  Week 72 (n=30, 19) | -0.2 (0.11) | 0.1 (0.07)

22. Secondary Outcome: Percentage of Participants With Beck Depression Inventory Fast Screen (BDI-FS) Score ≥ 4 at Each Time Point Assessed
Description: The BDI-FS consisted of seven areas with four statements (labeled 0, 1, 2, and 3) offered to describe the area of interest, with 0 indicating no effect and 3 indicating the worst effect. The individual area scores were summed to provide a total score. The degree of depression was assessed with 0 to 3 indicating minimal depression, 4 to 8 mild depression, 9 to 12 moderate depression and 13 to 21 severe depression.
Time Frame: Weeks 4, 8,12,16,20,24,28,32,36,40,44,48,60,72
Population: Participants from the Safety population who received at least one dose of study drug and who had data available at the given time point for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Number analyzed (Participants) | 77 | 75
Percentage of Participants
  Week 4 (n=61, 71) | 6.6 | 12.7
  Week 8 (n=57, 69) | 5.3 | 7.2
  Week 12 (n=55, 67) | 10.9 | 11.9
  Week 16 (n=50, 62) | 6.0 | 4.8
  Week 20 (n=46, 59) | 8.7 | 3.4
  Week 24 (n=45, 60) | 2.2 | 10.0
  Week 28 (n=46, 59) | 8.7 | 3.4
  Week 32 (n=37, 46) | 5.4 | 4.3
  Week 36 (n=37, 46) | 5.4 | 6.5
  Week 40 (n=42, 44) | 4.8 | 2.3
  Week 44 (n=36, 40) | 0 | 2.5
  Week 48 (n=32, 45) | 0 | 0
  Week 60 (n=1, 3) | 0 | 33.3
  Week 72 (n=30, 39) | 3.3 | 7.7

ADVERSE EVENTS:
Time Frame: 72 weeks for those patients who participated in the 48 week anti-HCV treatment period and the 24 week follow-up period plus an additional 16 weeks for those participants in the arm that received pioglitazone for 16 weeks during the run-in period.
Description: Safety population includes participants who received at least one dose of study drug and who had at least one post baseline safety assessment.
Arm/Group | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone | PEG-INF Alpha-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 10/77 | 9/75
Other Adverse Events (participants affected / at risk) | 68/77 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone (N=77) | PEG-INF Alpha-2a + Ribavirin (N=75)
Pneumonia (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-INF Alpha-2a + Ribavirin+ Pioglitazone (N=77) | PEG-INF Alpha-2a + Ribavirin (N=75)
Fatigue (General disorders) | 30 | 35
Influenza like illness (General disorders) | 13 | 12
Pyrexia (General disorders) | 12 | 7
Injection site erythema (General disorders) | 1 | 17
Irritability (General disorders) | 8 | 7
Pain (General disorders) | 12 | 3
Chills (General disorders) | 6 | 5
Injection site reaction (General disorders) | 1 | 6
Oedema peripheral (General disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 26 | 21
Diarrhoea (Gastrointestinal disorders) | 9 | 10
Vomiting (Gastrointestinal disorders) | 6 | 9
Constipation (Gastrointestinal disorders) | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 6
Haemorrhoids (Gastrointestinal disorders) | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Toothache (Gastrointestinal disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 11 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 27 | 24
Neutropenia (Blood and lymphatic system disorders) | 15 | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 21 | 23
Depression (Psychiatric disorders) | 9 | 23
Anxiety (Psychiatric disorders) | 2 | 9
Suicidal ideation (Psychiatric disorders) | 5 | 0
Headache (Nervous system disorders) | 14 | 20
Dizziness (Nervous system disorders) | 12 | 12
Dysgeusia (Nervous system disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 5
Urinary tract infection (Infections and infestations) | 6 | 2
Bronchitis (Infections and infestations) | 6 | 1
Nasopharyngitis (Infections and infestations) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Weight decreased (Investigations) | 3 | 8
Weight increased (Investigations) | 4 | 0
White blood cell count decreased (Investigations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 8
Vision blurred (Eye disorders) | 4 | 5
Hypertension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.